CLINICAL TRIAL: NCT07077616
Title: Clinical Study for the Therapeutic Efficacy and Safety of a Personalized and AI-Quantum Mechanics Based and Molecular Modeled Cancer Specific Neoantigenic Vaccine, the TamavaqTM NeoVaccine in Patients With Newly Diagnosed Glioma.
Brief Title: Clinical Study for the Safety and Therapeutic Efficacy of the AI-QMMM Designed TamavaqTM Personalised Vaccine in Patients With Newly Diagnosed Glioma.
Acronym: TAMAVAQTM
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Biogenea Pharmaceuticals Ltd. (Industry)
Collaborators: Naval Hospital, Athens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Biogenea1; Biogenea1979 (Other: Biogenea)
Record Dates: First submitted 2025-06-18; First posted 2025-07-22 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-09

CONDITIONS: Glioma
Keywords: Personalised Vaccine; Neoantigenic Peptides; AI-designed; Machine Learning-predicted; Quantum Mechanics structured; Molecular Dynamics-modeled; Immunodominant Peptides
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Intervention Model Description: The study intervention for this AI-QMMM designed and glioma treated personalized neoantigenic vaccine clinical trial involves the administration of a customized vaccine designed to elicit a targeted immune response against specific neoantigens present in the participant's tumor. The TAMAVAQ's intervention aims to enhance the body's immune response to glioma cells, potentially improving clinical outcomes in patients with this challenging form of brain cancer. Collectively, our findings are going to suggest that TAMAVAQ can stimulated the expansion of neoantigen-specific effector T cells and provide encouraging results to aid in the development of future neoantigen vaccine-based clinical trials in patients with GBM. By combining personalized neoantigen identification with a robust vaccine platform and thorough immune monitoring, the TAMAVAQ trial aims to provide valuable insights into the safety and efficacy of this innovative treatment strategy in glioma patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: personalized vaccine patients with recurrent malignant gliomas enrolled into this arm (Experimental): Clinical event timeline and Dosing of TAMAVAQ VACCINES
  Clinical event timeline for the patients who received at least one vaccine dose of (20-200)μg TAMAVAQ NeoVaccine, will be calculated from surgery until time of death due to progressive disease. Median progression-free survival (PFS) and overall survival (OS) will be also calculated respectively. Among enrolled patients, a median of (110-145) somatic single-nucleotide variants per tumour (range, 75-158) will be tested with a median of (58-63) coding mutations per tumour (range, 32-93) using whole-exome sequencing, and the expression of a subset of genes will be confirmed by RNA sequencing (RNA-seq) analysis. These included mutations commonly observed in glioblastoma that affect PTEN, RB1 and EGFR. No IDH1 or IDH2 mutations will be also tested. A median of 60.5-70,8 HLA binders (range, 30-163) with a half-maximum inhibitory concentration (IC50) < 500 nM will be predicted per tumour.
  Interventions: Biological: Biological: personalized vaccine Based on genetic and transcriptional sequencing information, personalized peptide vaccines would be designed and produced;

INTERVENTIONS:
Biological: Biological: personalized vaccine Based on genetic and transcriptional sequencing information, personalized peptide vaccines would be designed and produced; — TAMAVAQ Vaccine plus Poly-ICLC, cGAMP, Granulocyte-macrophage colony stimulating factor (GM-CSF), imiquimod, CpG oligodeoxynucleotides, saponins and monophosphoryl lipid A (MPLA)
  * TAMAVAQ VACCINE : Each one of our TAMAVAQ VACCINE is consisted of 1-35 (LIMPs, ASPs, and bEPTs) Personalised Synthetic Neoantigenic Peptides mixed with GBM TAAs, including MAGE-1, HER-2, gp100, AIM-2, TRP-2, EphA2,105 survivin50, IL13Rα2, heat-shock peptide protein complex-96 (HSPPC-96), and Smac-TLR7/8 peptides.
  * TAMAVAQ vaccine products are composed of 1-35 peptides from the Biogenea Pharmaceuticals Ltd warehouse.
  * TAMAVAQ vaccine will be applied before maintenance TMZ cycles after completion of chemoradiation therapy (CRT). Beginning on day 14 before the first maintenance TMZ cycle, patients will receive 7 vaccinations with TAMAVAC VACCINE

SUMMARY:
Gliomas are a heterogeneous group of tumors arising from glial cells in the central nervous system and are associated with poor prognosis and significant morbidity. The most aggressive form, glioblastoma multiforme (GBM), remains particularly challenging to treat, often exhibiting resistance to conventional therapies such as chemotherapy and radiation. The average survival for patients with GBM is approximately 15 months, underscoring the urgent need for novel therapeutic strategies that can improve outcomes. Malignant gliomas are the most common primary brain cancer diagnosed and still carry a poor prognosis despite aggressive multimodal management. Despite the continued advances in immunotherapy for other cancer types, however, there remain no FDA approved immunotherapies for cancers such as glioblastoma. Neoantigen vaccines are a form of immunotherapy involving the use of DNA, mRNA, and proteins derived from non-synonymous mutations identified in patient tumor tissue samples to stimulate tumor-specific T-cell reactivity leading to enhance tumor targeting. Up to and including the current time, we have only nascent understandings, at the molecular and submolecular level, of how immunity is generated and maintained. As a result, we do not have fundamental mechanistic understandings of vaccine:antigen interactions, of vaccine-directed and initiated routes of immunity, nor how, through adjuvants and changes in our biologic environment (such as the intestinal microbiome), we might direct such immune responses. In particular, in the field of vaccinology we have few collaborations between biology, physics, and chemistry...or what has been termed "convergence science"...but particularly from physics and the field of quantum mechanics. Biophysics led to quantum biology and quantum immunology reflecting quantum dynamics within living systems and their evolution. Unfortunately, despite the seismic influence of immunotherapy on oncology today, there remain no FDA approved immunotherapies for GBM due to the lack of efficacy observed in several randomized clinical trials. The TAMAVAQ approaches enable a quantitative understanding of immune response kinetics following neoantigen-based peptide vaccine treatment. Insights gained from challenges can be used to design better vaccines and evaluate the potential candidate vaccines in silico. The TAMAVAQ models also can guide such decisions on treatment regimens such as dosing and infusion frequencies.

DETAILED DESCRIPTION:
Quantum Vaccinomics for the Generation of the TAMAVAQ personalized neoantigenic vaccines.

The personalized neoantigen vaccines will be prepared based on the analysis of whole-exome sequencing (WES) and RNA-seq data generated from fresh-frozen tumours or tumours that will be available as formalin-fixed paraffin-embedded (FFPE) tissue, obtained at the time of diagnostic resection. WES of normal tissue will be generated from autologous PBMC DNA. Patient HLA allotype will be assessed using standard class I and class II PCR-based typing (BWH Tissue Typing Laboratory). Coding mutations will be identified and personal neoantigens will be predicted based on binding affinity analysis to individual HLA alleles using class I MHC binding prediction tools with a cut-off of predicted IC50 < 500 nM for selected epitopes. Quantum Circuit platforms for the identification of immunological quantum and design of TAMAVAQ's NeoVaccine consisted of Druggable Immunodominant and Immunogenic Neo-epitopic Peptides will be incorporated in this clinical study. Candidate and Prioritized Neo-epitopic Peptides are identified using systems biology integration of omics dataset combined with Big Data analytics and machine learning. Then, the immunodominant quantized peptide will be identified by using in silico algorithms and HLA epitope mapping and binding domains involved in each one Glioma Patient's Drug-DNA-Protein-protein interactions.

This clinical trial provides an AI-QMMM method for the identification and characterization of neoantigens and outlines the clinical applications of prospective immunotherapeutic strategies based on neoantigens exploring their current status, inherent challenges, and clinical translation potential against Glioma medical conditions.

Enhanced Targeted Therapy**:- The TAMAVAQ vaccine specifically targets neoantigens unique to glioma cells, potentially leading to a more effective immune response while sparing healthy cells. This specificity may reduce collateral damage associated with traditional cancer therapies.

Immune System Activation**:The TAMAVAQ personalized vaccine is designed to stimulate the patient's immune system, enhancing its ability to recognize and attack glioma cells. This activation can lead to a more robust and sustained anti-tumor response.

Potential for Long-term Remission**:- By training the immune system to identify and remember glioma cells, patients may achieve longer-lasting remission rates and a reduced likelihood of tumor recurrence compared to conventional therapies.**Reduction in Side Effects**:- Compared to traditional treatments such as chemotherapy and radiation, which often come with significant side effects, the TAMAVAQ personalized neoantigen vaccine may result in fewer adverse effects, thereby improving the patient's quality of life.

Personalized Treatment Approach**:- Each TAMAVAQ vaccine is tailored to the individual patient's tumor profile, potentially increasing the efficacy of the treatment. This personalization allows for a more precise approach to therapy that aligns with the unique characteristics of each Glioma patient's cancer.

Opportunities for Combination Therapies**:- The TAMAVAQ vaccine can potentially be used in conjunction with other treatments (e.g., checkpoint inhibitors, targeted therapies), enhancing overall treatment effectiveness and providing a multifaceted approach to combat glioma.**Real-time Monitoring and Adaptation**:- This clinical trial setting allows for continuous monitoring of patient responses, providing valuable data that can lead to adaptations in treatment strategies based on observed efficacy and safety profiles.

Contribution to Scientific Knowledge**:- The TAMAVAQ trial can provide critical insights into the mechanisms of immune responses against gliomas, contributing to the broader understanding of cancer immunotherapy and paving the way for future treatments.**Potential for Broader Application**:Success in the glioma trial may lead to the development of similar personalized vaccines for other cancer types, expanding the impact of this innovative therapeutic approach.**Patient Empowerment and Engagement**:Participation in TAMAVAQ clinical trials often empowers patients by involving them in cutting-edge research, providing them with access to novel therapies and fostering a sense of hope in their treatment journey.

This TAMAVAQ clinical trial holds substantial potential benefits, ranging from enhanced targeted therapy and immune activation to improved patient quality of life and contributions to scientific knowledge. As research progresses, it is essential to continue evaluating these benefits in conjunction with the associated risks to optimize treatment strategies for glioma patients.The development of the TAMAVAQ personalized vaccine represents a novel approach to glioma treatment. This analysis evaluates the potential risks and benefits associated with conducting a clinical trial for this innovative therapeutic strategy.

This clinical trial aims to assess the safety, tolerability, and efficacy of a personalized neoantigenic vaccine designed for patients diagnosed with glioma. The TAMAVAQ study will involve identifying patient-specific neoantigens from tumor biopsies and formulating tailored vaccines to stimulate an immune response against glioma cells. Following surgery, patients will receive conventional radiation therapy administered at 180-200 cGy per fraction daily for five days per week to a total of approximately 60 Gy. Personalized neoantigen vaccines TAMAVAQ NeoVaccine will be prepared using information from fresh tumour and normal tissue obtained at the time of diagnostic resection, as described below. Algorithms and methods based on profiles of sequence motifs, quantitative matrices (QM), artificial neural networks (ANN), support vector machines (SVM), quantitative structure activity relationship (QSAR), T-cell major histocompatibility complex (MHC) class I binding prediction and molecular docking simulations among others will be combined and used in order to predict and design the TAMAVAQ NeoVaccine-Drug Product Neo-epitopes. Quantum chemical calculations (IBM Quantum Studio) will be used to predict the TAMAVAQ NeoVaccine-Drug Product's biological function and be applied to T-cell receptor interaction with TAMAVAQ NeoVaccine-Drug Product Peptide/MHC class I. A cluster of algorithms is proposed here using semi-empirical quantum mechanical methods for calculating peptide-MHC class I and II molecules binding energy for the rational design of T-cell TAMAVAQ NeoVaccine-Drug Product Neo-epitopes with application in cancer glioma vaccinology. The vaccine will be administered subcutaneously at least seven to twelve weeks following completion of external beam radiotherapy. TAMAVAQ NeoVaccine-Drug Product will be applied before maintenance of TMZ cycles after completion of chemoradiation therapy (CRT). Beginning on day 14 before the first maintenance TMZ cycle, patients will receive 7 vaccinations with TAMAVAQ NeoVaccine drug products during 7 weeks. 20-200 μg per peptide per vial are used followed by two booster doses eight and sixteen weeks later. For each dose, vaccine will be administered within six hours of thawing in a non-rotating fashion to one of up to four extremities. Patients will be repeatedly vaccinated with TAMAVAQ NeoVaccine drug products beginning on day 33 of the 6 maintenance TMZ cycle. Patients will receive 9 vaccinations within 12 weeks. 20-400 μg per peptide per vial will be used. Concomitant medications deemed necessary for adequate patient care will be allowed, including concomitant corticosteroids for symptoms associated with cerebral oedema, but the study vaccine will be held for patients requiring more than 4 mg per day of dexamethasone within seven days of vaccine administration. Clinical assessment and monitoring will be delivered by using the RANO criteria and the Immunotherapy Response Assessment in the Neuro-Oncology criteria.

Study Design

* Type**: Open-label, single-arm, multicenter clinical trial
* Phase**: Phases I & II
* Duration**: Approximately 24 months (including recruitment, treatment, and follow-up) Methodology

Screening Phase (Month 1-2)**:

Recruitment**: Patients will be recruited from participating medical centers and clinics.

Informed Consent**: Obtain informed consent from eligible patients. Screening Assessments**: Conduct baseline assessments, including medical history, imaging, and laboratory tests to confirm eligibility.

Vaccine Development Phase (Month 3-5)**:

Tumor Biopsy**: Collect tumor samples from enrolled patients for sequencing and neoantigen identification.

Neoantigen Identification**: Utilize computational algorithms and laboratory techniques to identify patient-specific neoantigens.

Vaccine Formulation**: Develop personalized vaccines based on identified neoantigens tailored to each patient.

Vaccination Phase (Month 6)**:

-**Pre-Vaccination Assessments**: Conduct baseline assessments, including physical examinations and laboratory tests before vaccine administration.

* TAMAVAQ Vaccine Administration**: Administer the TAMAVAQ personalized neoantigenic vaccine via subcutaneous or intradermal injection.
* Immediate Post-Vaccination Monitoring**: Monitor patients for immediate side effects and adverse reactions for a specified period following vaccination.

Follow-Up Phase (Month 7-24)**:

Regular Follow-Up Visits**: Schedule follow-up visits at regular intervals (e.g., every 4-6 weeks) to assess patient health, side effects, and immune response.

Adverse Event Monitoring**: Continuously monitor and report any adverse events or serious adverse events to regulatory authorities.**Imaging and Laboratory Assessments**: Conduct imaging studies (e.g., MRI) and laboratory tests to evaluate treatment response and tumor status at designated follow-up intervals.

Quality of Life Assessments**: Administer validated quality of life questionnaires at baseline and follow-up visits to assess the impact of AI-QMMM designed TAMAVAQ treatment.**Study Closure (Month 24)**:

Final Patient Assessments**: Conduct final assessments for all participants to evaluate long-term outcomes and safety.

Data Analysis and Reporting**: Analyze TAMAVAQ trial data and prepare reports for submission to regulatory authorities and publication in scientific journals.

Feedback and Follow-Up**: Provide TAMAVAQ vaccinated participants with feedback on trial outcomes and offer continued follow-up care or access to alternative treatments as needed.

Sample Size - Estimated based on expected effect size and power calculations, aiming for a target enrollment of approximately 50-140 patients to provide adequate statistical power for the primary and secondary endpoints.

Statistical Analysis

Descriptive Statistics**: To summarize demographic and baseline characteristics.

Efficacy Analysis**: Kaplan-Meier survival curves for progression-free survival (PFS) and overall survival (OS).

Adverse Events Analysis**: Frequency and severity of adverse events reported according to NCI CTCAE criteria.

ELIGIBILITY:
Inclusion Criteria:

* 1. **Age**:
* Patients must be aged 18 years or older.
* signed inform consent;
* patients with recurrent malignant glioma; have received surgery, radiotherapy, chemotherapy;
* patients' tumor tissue should have a high mutation load(>10 TMB); be genetically unstable; at least have 10 neoantigens;
* should be able to provide tumor tissue and peripheral blood for sequencing and flow cytometry analysis;
* at least three months post last operation; one month after the completion of the last anti-drug therapy or radiotherapy;
* have not received any immunotherapy;
* at least have one measurable lesion;
* KPS >60;
* estimated survival > 3 months
* patients should have adequate organ and bone marrow function; 2. **Diagnosis**:
* Histologically confirmed diagnosis of glioma, including:
* Glioblastoma multiforme (GBM, WHO grade IV)
* Anaplastic astrocytoma (WHO grade III)
* Diffuse astrocytoma (WHO grade II)
* Other gliomas (e.g., oligodendroglioma, mixed glioma) confirmed by pathology.

  3. **Measurable Disease**:
* Presence of measurable disease, defined as at least one tumor lesion that can be accurately assessed by imaging techniques (e.g., MRI) according to RECIST criteria.

  4. **Performance Status**:
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2, indicating that patients are fully active, restricted in physically strenuous activity, or unable to work but able to care for themselves.

  5. **Adequate Organ Function**:
* Laboratory results must indicate adequate organ function, including:
* Hematological parameters: Hemoglobin ≥ 9 g/dL, white blood cell count ≥ 3,000 cells/mm³, platelet count ≥ 100,000 cells/mm³.
* Liver function tests: Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels ≤ 2.5 times the upper limit of normal (ULN) (or ≤ 5 times the ULN if there is liver involvement).
* Renal function: Serum creatinine ≤ 1.5 times the ULN or estimated glomerular filtration rate (eGFR) ≥ 60 mL/min.

  6. **Informed Consent**:
* Provision of written informed consent by the patient or their legally authorized representative, indicating understanding of the study procedures, potential risks, and benefits.

  7. **No Prior Treatment with Certain Therapies**:
* Patients must not have received prior treatment with immune checkpoint inhibitors or other experimental immunotherapies that may interfere with the study outcomes.

  8. **Ability to Comply with Study Procedures**:
* Patients must be able to comply with all study procedures, including follow-up visits and assessments, as determined by the investigator.

  9. **No Significant Cognitive Impairment**:
* Patients must not have significant cognitive impairment or psychiatric disorders that would compromise their ability to provide informed consent or adhere to the study protocol.

These inclusion criteria are designed to ensure that the study population for this glioma targeted personalized neoantigen vaccine clinical trial is suitable for participation, allowing for the collection of meaningful data regarding the safety and efficacy of the investigational treatment. By clearly defining eligibility, the trial aims to target patients who are most likely to benefit from this AI-QMMM inspired therapeutic approach.

Exclusion Criteria: 1. **Previous Treatments**:

* Patients who have received prior treatment with immune checkpoint inhibitors, other cancer vaccines, or experimental immunotherapies that may interfere with the study outcomes.

  2. **Active Autoimmune Diseases**:
* Patients with active autoimmune diseases or chronic inflammatory conditions requiring systemic treatment (e.g., rheumatoid arthritis, lupus, multiple sclerosis).

  3. **Pregnancy or Breastfeeding**:
* Pregnant or breastfeeding women, as the effects of the vaccine on fetal development or breastfeeding infants are not yet established.

  4. **Other Malignancies**:
* Patients with any other malignancy within the past 5 years, except for non-melanoma skin cancer or localized prostate cancer that is not currently active.

  5. **Uncontrolled Medical Conditions**:
* Patients with uncontrolled medical conditions, including but not limited to:
* Cardiovascular disease (e.g., recent myocardial infarction, severe heart failure).
* Uncontrolled infections (e.g., HIV, active hepatitis B or C).
* Severe chronic lung disease.

  6. **Significant Cognitive Impairment**:
* Patients with significant cognitive impairment or psychiatric disorders that would limit their ability to provide informed consent or comply with study procedures.

  7. **Severe Allergies**:
* Patients with known hypersensitivity or severe allergic reactions to any component of the vaccine formulation or adjuvants used in the study.

  8. **Concurrent Participation in Other Clinical Trials**:
* Patients currently participating in other clinical trials involving investigational drugs or therapies that may interfere with the study outcomes.

  9. **History of Organ Transplant**:
* Patients who have received an organ transplant that requires ongoing immunosuppressive therapy.

  10. **Severe Comorbidities**:
* Patients with severe comorbid conditions that, in the opinion of the investigator, may compromise the safety of the patient or interfere with the assessment of the study endpoints. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
TAMAVAQ Vaccine Safety Analysis | From initiation of study treatment to 28 weeks post-vaccination
  The primary objective of this study is to determine the safety of TAMAVAQ in patients with glioblastoma and to determine if TAMAVAQ shows sufficient safety in these patients. The safety assessments outlined for the TAMAVAQ vaccine clinical trial are essential for ensuring participant well-being and monitoring the impact of the intervention. The primary outcomes assessed by this clinical study were safety and efficacy of the TAMAVAQ autologous neoantigenic vaccine products based on reported adverse events (AEs) and clinical response respectively. To evaluate the safety of a neoantigen cancer vaccine, the Investigators monitor for adverse events using standardized criteria like the Common Terminology Criteria for Adverse Events (CTCAE) and assess changes in blood, urine, and organ function. They also track health-related quality of life.The Investigators will use the CTCAE to grade and track adverse events (side effects) that occur during and after TAMAVAQ vaccination.
Incidences of Advent Events and Severe Advent Events | From initiation of study treatment to 28 weeks post-vaccination
  Safety oversight is a critical component of clinical trials, ensuring that participant safety is prioritized throughout the study. Below is an outline of the safety oversight mechanisms and procedures for an AI and quantum mechanics-based brain tumor targeted personalized neoantigenic peptide vaccine clinical trial.
  * The safety of the TAMAVAQ vaccines will be evaluated by analyzing the rate of Grade 1-3 Treatment Related Adverse Events (TRAEs). The specific adverse events to be monitored include:
  * **Fever**
  * **Headache**
  * **Flu-like Symptoms**
  * **Lymphopenia**
  * **Injection Site Reactions**
  * **Vomiting**
  * **Diarrhea**
  * By systematically reviewing data from multiple studies, the analysis aims to quantify the incidence of these adverse events and provide a comprehensive understanding of the TAMAVAQ vaccine's safety profile.This provides a standardized way to assess the severity and frequency of potential safety issues.
Physiological Monitoring and Toxicity Analysis | From initiation of study treatment to 28 weeks post-vaccination
  Physiological Monitoring: Changes in blood counts, urine analysis, liver and kidney function tests, and electrolyte and coagulation parameters are monitored before and after TAMAVAQ vaccination to detect any physiological abnormalities that could be related to the TAMAVAQ vaccine. This structured approach enhances the reliability of trial outcomes and contributes to the advancement of the TAMAVAQ personalized cancer therapies for glioma patients. Toxicity Analysis: The Investigators will evaluate the overall toxicity profile of the vaccine, considering the frequency and severity of adverse events.
Gadolinium-enhanced MRI | From initiation of study treatment to 28 weeks post-vaccination
  To evaluate the safety of the TAMAVAQ neoantigen vaccines in glioma patients using Gadolinium-enhanced MRI, the primary approach involves monitoring changes in tumor size and characteristics over time, specifically using the McDonald criteria. These criteria, applied to gadolinium (Gd)-enhanced T1-weighted images, assess tumor response based on the appearance of the pre-treatment MRI. Additionally, T2-weighted images and potentially other advanced MRI techniques like dynamic susceptibility contrast (DSC)-MRI will provide further insights into tumor progression, pseudoprogression, and immune activity. Gadolinium-enhanced T1-weighted images: These images are crucial for visualizing areas of increased vascular permeability, which often indicate tumor growth or recurrence.
AI Techniques and Machine Learning Models for the TAMAVAQ's Safety Integration Analysis | From initiation of study treatment to 28 weeks post-vaccination
  Data Cleansing & Normalization: Handling heterogeneous data formats. Consider incorporating machine learning algorithms to improve the safety of the TAMAVAQ's vaccine neoantigen prediction and patient stratification based on historical data.
  * **Natural Language Processing (NLP):** Extract insights from unstructured clinical notes, glioma pathology reports.
  * **Machine Learning Models:**
  * Supervised learning for predicting TAMAVAQ's treatment safety outcomes.
  * Unsupervised clustering for TAMAVAQ's patient stratification.
  * **Predictive Modeling:** Identifying unstructured factors associated with TAMAVAQ's safety.
  * **Meta-Analytic Framework:** Combining effect sizes across studies to derive overall estimates.
  * Safety profile comparison with other Glioma targeted immunotherapies.

SECONDARY OUTCOMES:
Revised Assessment in Neuro-Oncology (RANO) Criteria for measuring the effectiveness of TAMAVAQ treatments in glioma patients. | From initiation of study treatment to 48 weeks post-vaccination
  The RANO (Response Assessment in Neuro-Oncology) criteria will be used to evaluate the effectiveness of TAMAVAQ treatments for glioma patients by assessing changes in tumor size and neurological function. RANO relies on MRI scans to measure tumor dimensions and considers both enhancing and non-enhancing tumor components. Clinical assessments, including neurological status and steroid use, will also be integrated into the evaluation, after TAMAVAQ treatment indicating whether the tumor is responding to TAMAVAQ's vaccine therapy.
Measurable Lesions and Macdonald Criteria | From initiation of study treatment to 48 weeks post-vaccination
  Measurable Lesions: Defined as contrast-enhancing or non-contrast-enhancing lesions with clear margins on MRI and perpendicular diameters of at least 10 mm.
  Response Categories:
  Complete Response (CR): Disappearance of all measurable lesions. Partial Response (PR): At least a 50% decrease in the sum of the products of perpendicular diameters of measurable lesions, sustained for at least 4 weeks.
  Stable Disease (SD): Neither sufficient decrease to qualify as PR nor sufficient increase to qualify as PD.
  Progressive Disease (PD): At least a 25% increase in the sum of the products of perpendicular diameters of measurable lesions or the appearance of new lesions. The MacDonald criteria will be used to assess treatment response in the TAMAVAQ vaccinated glioma patients by evaluating changes in tumor size on MRI scans alongside clinical assessment and corticosteroid use.
MRI Advanced Imaging Techniques | From initiation of study treatment to 48 weeks post-vaccination
  MRI (Magnetic Resonance Imaging) is an essential tool in evaluating brain tumors, and the use of advanced sequences significantly enhances its diagnostic capabilities. In the context of TAMAVAQ vaccinated patients, these advanced MRI techniques can provide valuable information about tumor characteristics. Advanced imaging techniques like MRI scans will play a crucial role in assessing the clinical efficacy of the TAMAVAQ treatments by providing detailed information about tumor characteristics, TAMAVAQ vaccine treatment response, and potential recurrence. These techniques will help in grading gliomas, distinguishing between TAMAVAQ treatment effects and tumor progression, and optimizing TAMAVAQ vaccine treatment strategies.
Perfusion Imaging (DSC, DCE, ASL) | From initiation of study treatment to 48 weeks post-vaccination
  Dynamic Susceptibility Contrast (DSC) and Dynamic Contrast-Enhanced (DCE) imaging assess tumor vascularity and blood flow will help to understand the tumor's angiogenesis and TAMAVAQ's treatment response.
  Arterial Spin Labeling (ASL) is a non-invasive method that measures cerebral blood flow without the need for contrast agents, which can be particularly beneficial in monitoring patients post-TAMAVAQ vaccinations.
Diffusion Imaging (DTI, DKI) | From initiation of study treatment to 48 weeks post-vaccination.
  Diffusion Tensor Imaging (DTI) and Diffusion Kurtosis Imaging (DKI) provide insights into tissue cellularity and microstructural integrity. These techniques will help differentiate between viable tumor tissue and areas of necrosis or edema after TAMAVAQ treatment indicating whether the tumor remains viable to TAMAVAQ's vaccine therapy. In the context of TAMAVAQ treatment, employing DTI and DKI can be instrumental in monitoring therapeutic efficacy. By analyzing these parameters, the investigators will differentiate between residual viable tumor tissue and non-viable areas post-treatment, aiding in the assessment of whether the tumor remains active and responsive to the Cancer Specific Neoantigenic TAMAVAQ vaccine therapy.
Magnetic Resonance Spectroscopy (MRS) | From initiation of study treatment to 48 weeks post-vaccination.
  Magnetic Resonance Spectroscopy (MRS) will offer metabolic information by analyzing the concentrations of specific metabolites within the tumor, which can indicate tumor aggressiveness and response to TAMAVAQ treatment. MRS will detect during and after TAMAVAQ vaccinations a wide range of metabolites, including: N-acetylaspartate (NAA): A marker of neuronal health and function, Creatine (Cr): An indicator of cellular energy metabolism, Choline (Cho): A marker of cell membrane turnover and proliferation, Myo-inositol (mI): A marker of glial cell activity, Lactate (Lac): An indicator of anaerobic metabolism, and Glutamate/Glutamine (Glx): Neurotransmitters.
PET Advanced Imaging Techniques: PET scans | From initiation of study treatment to 48 weeks post-vaccination.
  PET scans, using tracers like FET or FLT, will be used to assess tumor metabolism and proliferation, providing information about tumor activity and response to TAMAVAQ therapy.
  FET-PET: FET-PET will help delineate the extent of the tumor, especially in areas not visible on MRI, and will be used to guide radiation therapy planning in TAMAVAQ vaccinated patients: FET-PET (Fluoroethyltyrosine Positron Emission Tomography) is indeed a valuable imaging tool in oncology, particularly for brain tumors.In the context of TAMAVAQ vaccinated patients, using FET-PET can enhance the understanding of tumor behavior post-vaccination, as it helps in assessing the tumor's response to the therapy and adjusting treatment plans accordingly. This approach can lead to more targeted and effective TAMAVAQ vaccination therapy, potentially improving patient outcomes.
Diffusion-weighted Images (DWI) | From initiation of study treatment to 48 weeks post-vaccination.
  Diffusion-weighted Images (DWI): Diffusion-weighted imaging (DWI) in glioma patients participating in the TAMAVAQ clinical trial is a powerful tool for assessing tumor characteristics and TAMAVAQ treatment response. It will measure water molecule movement, reflecting tissue cellularity and microstructure, which will be used to track tumor progression, and evaluate TAMAVAQ therapy effectiveness. DWI will be used to assess clinical efficacy in TAMAVAQ vaccinated glioma patients.
DWI for Monitoring TAMAVAQ's Treatment Responses | From initiation of study treatment to 48 weeks post-vaccination.
  Pre-treatment Assessment: DWI will determine the baseline characteristics of the tumor before TAMAVAQ treatment, providing a benchmark for comparison with post-TAMAVAQ-treatment scans. DWI will generate ADC maps, which quantify water diffusion. Lower ADC values indicate restricted diffusion, often associated with higher tumor cell density and malignancy.
  Early Response Assessment: Changes in ADC values after TAMAVAQ treatment will indicate whether the tumor is responding to therapy. For example, an increase in ADC values may suggest a decrease in tumor cellularity due to TAMAVAQ treatment.
DWI for Assessing Tumor Infiltration and Recurrence for Standard DWI Protocols and Analysis | From initiation of study treatment to 48 weeks post-vaccination.
  Peritumoral Tissue Assessment:
  DWI will help to identify areas of tumor infiltration into surrounding brain tissue, even when these areas are not visible on conventional MRI, after TAMAVAQ treatment indicating whether the tumor is responding to TAMAVAQ vaccine therapy.
  Recurrence Detection:
  DWI will aid in the detection of tumor recurrence by identifying areas of restricted diffusion that may indicate tumor regrowth, after TAMAVAQ treatment indicating whether the tumor is responding to TAMAVAQ vaccine therapy.
  b-values: DWI is typically acquired with multiple b-values (e.g., 0, 1000 s/mm2) to calculate ADC values.
  Regions of Interest (ROIs):
  ROIs are placed on the tumor and surrounding normal-appearing white matter to obtain ADC measurements, after TAMAVAQ treatment indicating whether the tumor is responding to TAMAVAQ vaccine therapy.
Diffusion-tensor Imaging (DTI) for Monitoring TAMAVAQ's Treatment Responses | From initiation of study treatment to 48 weeks post-vaccination.
  Diffusion-tensor Imaging (DTI): Diffusion Tensor Imaging (DTI) is a valuable tool for assessing the clinical efficacy in the glioma patients participating in the TAMAVAQ clinical Trial by providing insights into tumor characteristics and TAMAVAQ treatment response. DTI measures the diffusion of water molecules within tissues, which is affected by the tissue's microstructure. In the TAMAVAQ clinical trial, DTI will help to determine tumor grade, assess infiltration, and evaluate response to TAMAVAQ therapy. By tracking changes in DTI metrics over time, TAMAVAQ's clinical trial investigators and clinicians can assess whether the TAMAVAQ treatment is effective and make adjustments to the treatment plan as needed.
Circulating Tumor Cells (CTCs) | From initiation of study treatment to 48 weeks post-vaccination.
  Circulating Tumor Cells (CTCs): To assess the clinical efficacy of circulating tumor cells (CTCs) in TAMAVAQ vaccinated glioma patients, several approaches will be employed, including monitoring CTC counts over time, analyzing CTC characteristics (like expression of specific markers), and correlating CTC data with clinical outcomes. These methods aim to evaluate the presence, abundance, and behavior of CTCs as indicators of disease progression, TAMAVAQ treatment response, and overall prognosis.
Circulating Tumor DNA (ctDNA) | From initiation of study treatment to 48 weeks post-vaccination.
  Circulating Tumor DNA (ctDNA): ctDNA, fragments of tumor DNA circulating in the bloodstream, is a key biomarker. Techniques like NGS and ddPCR will identify mutations, copy number variations, and other genetic changes in before and after TAMAVAQ's vaccinations.ctDNA of the TAMAVAQ's clinical trial participants receiving the TAMAVAQ individualized neoantigen-directed immunotherapy will be monitored longitudinally, up to two years, using a unique hybrid next generation sequencing assay targeting tumor-informed and tumor-naïve variants. Patient-specific panels will be designed targeting an average of 144 variants per patient. A tumor-naïve universal panel will also be designed for inclusion with patient-specific panels to monitor recurrently mutated tumor hotspots (e.g., KRAS and TP53) and genes implicated in TAMAVAQ immunotherapy resistance (B2M, TAP1/2).
Genomic Alterations, Molecular Analysis, and Glioma Circulating Biomarkers in Liquid Biopsies | From initiation of study treatment to 48 weeks post-vaccination.
  Genomic Alterations: NGS panels 30 genes of known relevance for CNS tumors to detect mutations (ie, point mutations and small insertion/deletions) and analyze multiple genes simultaneously, identifying various genomic alterations such as single nucleotide polymorphisms (SNPs), small insertions and deletions (indels), copy number alterations (CNAs), and gene fusions during and after TAMAVAQ's vaccinations.
  Molecular Analysis & Liquid biopsy: Analyzing circulating tumor cells, exosomes, or other circulating biomarkers (GFAP (Glial Fibrillary Acidic Protein), YKL-40, EGFR (Epidermal Growth Factor Receptor), PTEN, S100A8, c-MYC, CD133, CD44, A2B5, CD15, CD171, IDH mutation status and 1p/19q codeletion, MGMT (O6-methylguanine-DNA methyltransferase) promoter methylation, H3F3A alterations, and ATRX gene mutations) in blood samples will provide information about the tumor microenvironment during and after TAMAVAQ's vaccination scheme.
High-throughput Gene Expression Profiling Analysis | From initiation of study treatment to 48 weeks post-vaccination.
  Gene Expression Profiles: To assess the clinical efficacy of gene expression profiles in TAMAVAQ vaccinated glioma patients, the investigators will analyze gene expression data from tumor samples, correlating it with clinical outcomes like survival and TAMAVAQ treatment response. This involves identifying gene expression signatures, patterns of gene expression associated with specific traits or outcomes, and validating these signatures in independent patient cohorts. Statistical methods, including survival analysis and machine learning, will then employed to assess the predictive power of these signatures.Mutations in the isocitrate dehydrogenase (IDH) genes are critical for glioma classification and prognosis. Techniques like real-time PCR and NGS are commonly used to detect IDH mutations.
  Other Key Genes:
  Besides IDH, other genes like ATRX, TP53, TERT, PTEN, EGFR, and CIC are frequently mutated in different glioma types and should be assessed.
TME Microenvironment Proteomic analysis | From initiation of study treatment to 48 weeks post-vaccination.
  Tumor Microenvironment: To assess the clinical efficacy of TAMAVAQ treatments targeting the tumor microenvironment (TME) in the TAMAVAQ's vaccinated glioma patients, the investigators will analyze various factors including the microenvironment's composition, immune cell infiltration, and the impact on tumor behavior. This involves a combination of imaging techniques, molecular analyses of tumor and surrounding tissue, and assessment of patient outcomes.
  Proteomic analysis: Several proteins have been identified as potential biomarkers for glioma, including GFAP, YKL-40, EGFR, and PTEN. These proteins will be used to help diagnose, classify, and potentially predict the response to TAMAVAQ treatment in glioma patients. Analyzing protein expression in tumor samples will provide insights into the cellular and molecular composition of the TME for real-time assessment of the tumor microenvironment during and after TAMAVAQ vaccinations.
Methylation Patterns | From initiation of study treatment to 48 weeks post-vaccination.
  Methylation Patterns: To assess the clinical efficacy of methylation patterns in the TAMAVAQ's treated patients, the investigators will analyze DNA methylation profiles using techniques like bisulfite sequencing, methylation-specific PCR (MSP), or microarray-based assays. These profiles will then be correlated with patient outcomes (survival, recurrence) and TAMAVAQ's treatment responses (e.g., to chemotherapy). Statistical methods like Kaplan-Meier analysis and log-rank tests will be used to compare survival differences between groups with distinct methylation patterns.
Immune T Cell Analysis in Glioma-Associated Microglia/Macrophages (GAMs) | From initiation of study treatment to 48 weeks post-vaccination.
  Flow cytometry and immunohistochemistry: These techniques can be used to identify and quantify different immune cell populations within the tumor microenvironment.
  Analysis of immune cell markers: Assessing the expression of specific immune cell markers can provide information about the immune response to TAMAVAQ's vaccination treatments.
  Glioma-Associated Microglia/Macrophages (GAMs):
  Gliomas contain immune cells, including GAMs, which play a complex role in tumor progression. Flow cytometry will help to identify and characterize these cells, including their levels of CD45 and CD11b expression during and after TAMAVAQ vaccinations.
  T Cell Analysis:
  Flow cytometry will analyze T cell populations (CD4+ and CD8+) in gliomas, including their activation status and cytokine production (like IFN-γ), which can be relevant to understanding immune responses and TAMAVAQ treatment responses.
Assessment of Tumor Behavior | From initiation of study treatment to 48 weeks post-vaccination.
  Tumor volume and growth rate: Tracking changes in tumor size and growth rate using imaging techniques or other methods can indicate treatment response.
  Invasion and metastasis: Analyzing the extent of tumor invasion and metastasis can provide information about TAMAVAQ's treatment efficacy.
Machine learning algorithms for Bioinformatics, Neoantigenic Predictions, and Computational Modeling | From initiation of study treatment to 48 weeks post-vaccination.
  Machine learning algorithms: These will be used to integrate data from different sources (imaging, molecular analysis, clinical data) to predict the TAMAVAQ's treatment response and identify potential therapeutic Glioma neoantigenic targets.This analysis will reveal patterns of gene expression associated with different TME subtypes and predict TAMAVAQ's patient outcomes.
Survival Analysis | From initiation of study treatment to 48 weeks post-vaccination.
  In summary, measuring overall survival in glioma patients receiving neoantigen vaccines involves tracking patient survival times, generating survival curves, and analyzing the data statistically to assess the impact of the TAMAVAQ vaccine. This will be done in conjunction with monitoring the immune response to the TAMAVAQ vaccine to better understand how it may be affecting patient outcomes. Overall survival (OS) in glioma patients vaccinated with the TAMAVAQ neoantigen vaccines will be measured by tracking the time from vaccination to death from any cause. Survival curves will be generated (often using the Kaplan-Meier method) to visualize the OS data.
Longitudinal Tracking | From initiation of study treatment to 48 weeks post-vaccination.
  To measure the clinical efficacy of longitudinal tracking in TAMAVAQ vaccinated patients, the investigators will assess the TAMAVAQ's treatment response and disease progression over time using a combination of imaging, clinical assessments, and potentially, biomarkers. This involves tracking tumor burden, neurological function, patient-reported outcomes, and potentially, molecular markers.
TAMAVAQ Neoantigen Vaccines and miRNA Changes | From initiation of study treatment to 48 weeks post-vaccination.
  TAMAVAQ Neoantigen vaccines, designed to stimulate the immune system to target specific mutations in cancer cells, can induce changes in miRNA expression. Monitoring these changes can provide insights into the vaccine's efficacy.
  miR-21: Consistently upregulated in gliomas, involved in promoting tumor cell survival and invasiveness, and will be implicated in resistance to TAMAVAQ therapy combined to radiotherapy.
  miR-15b: Low expression will be associated with increased survival in TAMAVAQ vaccinated glioma patients.
  miR-128: Serum levels will differentiate TAMAVAQ vaccinated glioma patients from controls.
  miR-210: A promising biomarker for monitoring the effectiveness of the TAMAVAQ neoantigen-based vaccine in glioma patients.
  miR-155: Act as both an oncogene and a tumor suppressor, potentially influencing immune responses. Will identify early signs of treatment resistance, as miR-155 can be indicators of tumor recurrence or progression.

OTHER OUTCOMES:
Patient-Reported Outcomes (PROs) | From initiation of study treatment to 48 weeks post-vaccination
  Quality of Life (QoL) Questionnaires:
  Tools like the EORTC QLQ-C30 and BN20, FACT-G and Br, and MDASI-BT will be used to assess various aspects of QoL, including physical, emotional, social, and cognitive functioning.
  Symptom Scales:
  TAMAVAQ's vaccinated Patients will be reported on the severity of symptoms like fatigue, pain, and nausea/vomiting, providing valuable information about TAMAVAQ's treatment impact.
Neurological Examination | From initiation of study treatment to 48 weeks post-vaccination
  The TAMAVAQ clinical trial's clinicians and investigators will assess the patient's neurological status, including motor and sensory function, reflexes, and cognitive abilities.
  Karnofsky Performance Status (KPS):
  This scale measures a patient's overall functional status and ability to perform daily activities.

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis G Grigoriadis, Pharmacist, Study Director — Myoncotherapy
Locations (1):
- Biogenea Pharmaceuticals Ltd, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://myoncotherapy.com/wp-content/uploads/2025/05/TAMAVAC-TM-CLINICAL-PROTOCOL-IGG.pdf